CLINICAL TRIAL: NCT05093855
Title: A Multicenter, Open-label, Phase II Study to Explore Efficacy and Safety of BDB-001 Injection in Subjects With Moderate to Severe Hidradenitis Suppurativa
Brief Title: Efficacy and Safety Study of BDB-001 Injection in Patients With Moderate to Severe Hidradenitis Suppurativa (HS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Staidson (Beijing) Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STS-BDB001-08
Record Dates: First submitted 2021-06-23; First posted 2021-10-26 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — BDB001

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental)
  Interventions: Drug: BDB-001 Injection

INTERVENTIONS:
Drug: BDB-001 Injection — Multiple IV infusions of BDB-001 Injection diluted in sodium chloride

SUMMARY:
The purpose of this study is to explore whether BDB-001 Injection is effective and safe in the treatment of moderate to severe hidradenitis suppurativa(HS).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who signed the informed consent to participate in the STS-BDB001-06 clinical study and completed all follow-up of the study as required by the protocol, or who withdrew early due to treatment failure or other objective reasons and completed the early withdrawal visit (at least 4 weeks of treatment)

Exclusion Criteria:

* Never participated in the clinical study of STS-BDB001-06；
* Subjects withdrew from the STS-BDB001-06 clinical study due to an intolerable adverse event related to the study drug.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2023-08-22 (Actual); Study Completion 2023-08-22 (Actual)

PRIMARY OUTCOMES:
Change in International Hidradenitis Suppurativa Severity Score System (IHS4) score from Day 0 by time point | Week 8
  The International Hidradenitis Suppurativa Severity Score 4 (IHS4: developed by the European Hidradenitis Suppurativa Foundation Investigator Group)，IHS4 Score=(Nodule Count) + (Abscess Count*2) + (Draining Tunnel Count *4).
  IHS4 score uses a range grades:
  Mild=0-3; Moderate=4-10; Severe ≥11.

SECONDARY OUTCOMES:
Change in International Hidradenitis Suppurativa Severity Score System (IHS4) score from Day 0 by time point | From Day 0 until Day 56
  The International Hidradenitis Suppurativa Severity Score 4 (IHS4: developed by the European Hidradenitis Suppurativa Foundation Investigator Group)，IHS4 Score=(Nodule Count) + (Abscess Count*2) + (Draining Tunnel Count *4).
  IHS4 score uses a range grades:
  Mild=0-3; Moderate=4-10; Severe ≥11.
Change in modified Sartorius Score (mSS) from Day 0 by time point | From Day 0 until Day 56
  The mSS is a summation of HS lesions based on a number of factors including anatomical region, number and type of lesions, distance between relevant lesions and lesions clearly separated by normal skin in each region measured as HS clinical parameters. The scale title for mSS is points. The mSS has a minimum value of 0 and no upper limit. The higher the score the more severe is the disease/worse is the outcome.
Change in Hidradenitis Suppurativa Clinical Response (HiSCR) from Day 0 by time point | From Day 0 until Day 56
  The definition for response to treatment based on HiSCR relative to Baseline was: at least 50% reduction in abscesses and inflammatory nodule (AN) count (over all anatomical regions) with no increase in number of abscesses and in number of draining fistulas.
Change in Hidradenitis suppurativa-Physician Global Assessment (HS-PGA) score from Day 0 by time point | From Day 0 until Day 56
  Hidradenitis Suppurativa - Physician's Global Assessment (HS-PGA)classifies patients' severity into six categories:clear, minimal, mild, moderate, severe, and very severe, based on the number and quality of inflammatory lesions.
Changes of active lesions (number of inflammatory nodules, abscesses, fistulas, and abscess overflow score) from Day 0 by time point. | From Day 0 until Day 56
Change in Dermatology Life Quality Index (DLQI) score from Day 0 by time point | From Day 0 until Day 56
  A score is documented for each of the 10 DLQI items, ranging from 0 to 3 for each item. The scale title for DLQI is points. The total score is the sum of the responses to all 10 DLQI items, ranging from the minimum of 0 points to the maximum of 30 points. A higher score corresponds to worse health related quality of life/outcome.
7. Change in Dermatology visual analog scale (VAS) score from Day 0 by time point. | From Day 0 until Day 56]
Safety of BDB-001 injection in the treatment of patients with HS will be assessed | From Day 0 until Day 77
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Baoxi Wang, Master, Principal Investigator — Plastic Surgery Hospital,Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (15):
- China (15):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Plastic Surgery Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality
  - The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Union Hospital Tongji Medical College Huazong University of Science and Technology, Wuhan, Hubei
  - Xiangya Hospital, Central South University, Changsha, Hunan
  - Chinese Academy of Medical Sciences and Peking Union Medical College, Nanjing, Jiangsu
  - The First Hospital of Jilin Universitv, Changchun, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - The Second Affiliated Hospital of Air Force Medical University, Xi'an, Shaanxi
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Huashan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Skin Disease Hospital, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No